CLINICAL TRIAL: NCT07346066
Title: A Phase 3 Multi-Center Efficacy Study of Filricianine Injection in Patients Undergoing Robotic-Assisted Colorectal Surgery Using the da Vinci Surgical System With Firefly® Fluorescence Imaging
Brief Title: IS-001 Injection in Patients Undergoing Robotic-Assisted Colorectal Surgery
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Intuitive Surgical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ISI-124804-CR-3
Record Dates: First submitted 2026-01-14; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Ureter Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- IS-001 Injection (Other): Ureter visualization and delineation will be compared between white light (standard of care) and near-infrared (NIR) imaging mode after each of the two single intravenous injections of IS-001.
  Interventions: Drug: filricianine

INTERVENTIONS:
Drug: filricianine — IV injection of IS-001 filricianine with near infrared (NIR) imaging

SUMMARY:
This study evaluates the safety and efficacy of intravenous injection of IS-001 to aid in intraoperative ureter structure delineation

DETAILED DESCRIPTION:
Injury to the ureter, the duct by which urine passes from the kidney into the bladder, is a well-known and serious complication of pelvic and abdominal surgery that frequently goes unrecognized intraoperatively. This study seeks to evaluate the safety and efficacy of intravenous IS-001 injection to improve surgeon ureter visualization during robotic-assisted colorectal surgery with the da Vinci® Surgical System and Firefly® imaging.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female participants between the ages of 16 and 75, inclusive
2. Participant is scheduled to undergo robotic-assisted colectomy using the da Vinci X/Xi Surgical System with SFF Fluorescence Imaging Exclusion Criteria

1. Participant is pregnant or nursing 2. Participant has known current acute or chronic hepatitis B virus (HBV) or hepatitis C virus (HCV) infection 3. Participant has any of the following screening laboratory values: eGFR < 30 mL/min/1.73 m2

1. Aspartate aminotransferase (AST) ≥ 2.5 × ULN
2. Alanine aminotransferase (ALT) ≥ 2.5 × ULN
3. Total Bilirubin > 2mg/dL 4. Participant has any concomitant non-colorectal cancer 5. Participant has any circumstances that, in the judgment of the Investigator, might make them not a suitable candidate for the study 6. Participants have already been enrolled in another investigational drug or device study within the past 6 months 7. Participants with known or suspected hypersensitivity to indocyanine green (ICG) or any components of the formulation used 8. Participant is expected to receive or has received other methods for ureter identification during the surgery (e.g., ureteral stent placement, illuminated catheters, retrograde ICG injections) before the administration of IS-001 9. The duration of the surgery is expected to be less than 90 minutes as determined during preoperative planning.

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 146 (Estimated)
Dates: Start 2026-03-31 (Estimated); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Independent reader assessment of ureter visualization by 1-5 Likert visualization rating scale from 1 not visible, 2 questionably visible, 3 low visibility, 4 visible, 5 clearly visible. | 10 minutes after first injection
  Evaluate ureter visualization by each independent reader at (a) the pelvic brim (PB) and (b) Inferior Mesenteric Artery (IMA) locations in Sensitive Firefly (SFF) mode compared to white light mode up to 30 minutes after the first IS-001 injection.

SECONDARY OUTCOMES:
Independent reader assessment of ureter length delineation by line drawing on recorded frame measured in arbitrary unit length | 30 minutes after the first injection
  Evaluate ureter length delineation at (a) the PB and (b) IMA locations in SFF mode compared to white light mode up to 30 minutes after the first IS-001 injection
Independent reader assessment of ureter visualization by 1-5 Likert visualization rating scale from 1 not visible, 2 questionably visible, 3 low visibility, 4 visible, 5 clearly visible | 30 miinutes after second injection
  Evaluate ureter visualization by each independent reader at (a) PB and (b) IMA locations in SFF mode compared to white light mode up to 30 minutes after the second IS-001 injection
Independent reader assessment of ureter length delineation by line drawing on recorded frame measured in arbitrary unit length | 30 minutes after second injection
  Evaluate ureter length delineation at (a) the PB and (b) IMA locations in SFF mode compared to white light mode up to 30 minutes after the second IS-001 injection
Ureter visualization based on intraoperative surgeon's rating by 1-5 Likert visualization rating scale from 1 not visible, 2 questionably visible, 3 low visibility, 4 visible, 5 clearly visible | 30 minutes after first IS-001 injection
  Evaluate ureter visualization based on the intra-operative surgeon's rating at (a) the PB and (b) IMA locations in SFF mode compared to white light mode up to 30 minutes after the first IS-001 injection
Independent reader assessment of ureter visualization by 1-5 Likert visualization rating scale from 1 not visible, 2 questionably visible, 3 low visibility, 4 visible, 5 clearly visible. | 45 minutes after first injection
  Evaluate ureter visualization by each independent reader at (a) the PB and (b) IMA locations in SFF mode compared to white light mode up to 45 minutes after the first and second IS-001injection
Independent reader assessment of ureter visualization by 1-5 Likert visualization rating scale from 1 not visible, 2 questionably visible, 3 low visibility, 4 visible, 5 clearly visible | 45 minutes after second injection
  Evaluate ureter visualization by each independent reader at (a) the PB and (b) IMA locations in SFF mode compared to white light mode up to 45 minutes after the first and second IS-001injection
Concordance of ureter visualization between independent readers | 10 minutes after first injection
  Determine degree of concordance of ureter visualization between independent readers at (a) the pelvic brim and (b) the IMA location
Concordance of ureter visualization between independent readers | 30 minutes after first injection
  Determine degree of concordance of ureter visualization between independent readers at (a) the pelvic brim and (b) the IMA location
Concordance of ureter visualization between independent readers | 45 minutes after first injection
  Determine degree of concordance of ureter visualization between independent readers at (a) the pelvic brim and (b) the IMA location
Concordance of ureter visualization between independent readers | 10 minutes after second injection
  Determine degree of concordance of ureter visualization between independent readers at (a) the pelvic brim and (b) the IMA location
Concordance of ureter visualization between independent readers | 30 minutes after second injection
  Determine degree of concordance of ureter visualization between independent readers at (a) the pelvic brim and (b) the IMA location
Concordance of ureter visualization between independent readers | 45 minutes after second injection
  Determine degree of concordance of ureter visualization between independent readers at (a) the pelvic brim and (b) the IMA location
Concordance between intra-operative ureter visualization assessment and independent reader ureter visualization assessment | 10 minutes after first injection
  Determine the degree of concordance between the intra-operative ureter visualization assessment and the independent reader ureter visualization assessment
Concordance between intra-operative ureter visualization assessment and independent reader ureter visualization assessment | 30 minutes after first injection
  Determine the degree of concordance between the intra-operative ureter visualization assessment and the independent reader ureter visualization assessment
Concordance between intra-operative ureter visualization assessment and independent reader ureter visualization assessment | 45 minutes after first injection
  Determine the degree of concordance between the intra-operative ureter visualization assessment and the independent reader ureter visualization assessment
Concordance between intra-operative ureter visualization assessment and independent reader ureter visualization assessment | 10 minutes after second injection
  Determine the degree of concordance between the intra-operative ureter visualization assessment and the independent reader ureter visualization assessment
Concordance between intra-operative ureter visualization assessment and independent reader ureter visualization assessment | 30 minutes after second injection
  Determine the degree of concordance between the intra-operative ureter visualization assessment and the independent reader ureter visualization assessment
Concordance between intra-operative ureter visualization assessment and independent reader ureter visualization assessment | 45 minutes after second injection
  Determine the degree of concordance between the intra-operative ureter visualization assessment and the independent reader ureter visualization assessment
Degree of concordance of ureter visualization within independent readers | 10 minutes after first injection
  Determine degree of concordance of ureter visualization within independent readers at (a) the pelvic brim and (b) IMA location
Degree of concordance of ureter visualization within independent readers | 30 minutes after first injection
  Determine degree of concordance of ureter visualization within independent readers at (a) the pelvic brim and (b) IMA location
Degree of concordance of ureter visualization within independent readers | 45 minutes after first injection
  Determine degree of concordance of ureter visualization within independent readers at (a) the pelvic brim and (b) IMA location
Degree of concordance of ureter visualization within independent readers | 10 minutes after second injection
  Determine degree of concordance of ureter visualization within independent readers at (a) the pelvic brim and (b) IMA location
Degree of concordance of ureter visualization within independent readers | 30 minutes after second injection
  Determine degree of concordance of ureter visualization within independent readers at (a) the pelvic brim and (b) IMA location
Degree of concordance of ureter visualization within independent readers | 45 minutes after second injection
  Determine degree of concordance of ureter visualization within independent readers at (a) the pelvic brim and (b) IMA location
Ureter signal-to-background ratio evaluating contrast of fluorescent signal in NIR imaging mode | 10 minutes after first injection
  Evaluate ureter signal-to-background ratio in Firefly imaging at (a) the pelvic brim and (b) the IMA location
Ureter signal-to-background ratio evaluating contrast of fluorescent signal in NIR imaging mode | 30 minutes after first injection
  Evaluate ureter signal-to-background ratio in Firefly imaging at (a) the pelvic brim and (b) the IMA location
Ureter signal-to-background ratio evaluating contrast of fluorescent signal in NIR imaging mode | 45 minutes after first injection
  Evaluate ureter signal-to-background ratio in Firefly imaging at (a) the pelvic brim and (b) the IMA location
Ureter signal-to-background ratio evaluating contrast of fluorescent signal in NIR imaging mode | 10 minutes after second injection
  Evaluate ureter signal-to-background ratio in Firefly imaging at (a) the pelvic brim and (b) the IMA location
Ureter signal-to-background ratio evaluating contrast of fluorescent signal in NIR imaging mode | 30 minutes after second injection
  Evaluate ureter signal-to-background ratio in Firefly imaging at (a) the pelvic brim and (b) the IMA location
Ureter signal-to-background ratio evaluating contrast of fluorescent signal in NIR imaging mode | 45 minutes after second injection
  Evaluate ureter signal-to-background ratio in Firefly imaging at (a) the pelvic brim and (b) the IMA location

IPD SHARING:
Plan to Share IPD: No